CLINICAL TRIAL: NCT03759730
Title: Role of Microbiome as a Biomarkers in Locoregionally-Advanced Oropharyngeal Squamous Cell Carcinoma (ROMA LA-OPSCC)
Brief Title: Role of Microbiome as a Biomarkers in Locoregionally-Advanced Oropharyngeal Squamous Cell Carcinoma
Acronym: ROMA LA-OPSCC
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: ROMA LA-OPSCC-001
Record Dates: First submitted 2018-11-23; First posted 2018-11-30 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Locoregionally-advanced Oropharyngeal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, oropharyngeal swab over the tumor site, and stool sample are needed to assess the feasibility of microbiome evaluation in LA-OPSCC patients undergoing chemoradiotherapy (CRT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a minimal risk feasibility study involving the analysis of patient samples and does not involve any therapeutic intervention. The study will involve a prospective cohort of up to 60 patients diagnosed with Locoregionally-Advanced Oropharyngeal Squamous Cell Carcinoma (LA-OPSCC) treated with chemoradiotherapy (CRT) at Princess Margaret Cancer Centre.

DETAILED DESCRIPTION:
To assess the feasibility of microbiome evaluation in LA-OPSCC patients undergoing CRT using samples collected by four different methods: Saliva, Oropharyngeal swab over the tumor site (OP), Stool, and Rectal swab (optional).

This study is investigating the role of oral microbiota as a biomarker in LA-OPSCC. This is a minimal risk study involving the analysis of patient samples and does not involve therapeutic intervention. This protocol does not determine eligibility to receive treatment with concurrent radiotherapy and chemotherapy. It is anticipated that patient accrual will be completed within 12 months.

The study will involve a prospective cohort of up to 60 patients diagnosed with LA OPSCC treated with CRT at Princess Margaret Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written and voluntary informed consent.
2. Patient must be willing and able to provide collection for saliva, OP swab and stool specimen analyses at 2 time points. Rectal swab is optional.
3. Age > 18 years, male or female.
4. Patient must be diagnosed with histologically confirmed squamous cell carcinoma of the oropharynx (soft palate, tonsils, base of tongue).
5. Patients must be eligible for curative-intent concurrent treatment with radiotherapy and chemotherapy.

Exclusion Criteria:

- Any condition that, in the opinion of the Investigator, would interfere with patient safety, or evaluation of the collected specimen and interpretation of study result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with locoregionally-advanced oropharyngeal squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of microbiome evaluation in LA-OPSCC patients undergoing CRT using samples collected by four different methods | 1 year
  To assess the feasibility, the endpoint will be the proportion of analyzable samples.
Feasibility of microbiome evaluation in LA-OPSCC patients undergoing CRT using samples collected by four different methods | 1 year
  To assess the feasibility, the endpoint will be the patient compliance rate with sample collection timeline/procedures.

OTHER OUTCOMES:
Evaluation of the relationship between oral and intestinal microbiome composition and diversity in LA-OPSCC patients undergoing CRT. | 1 year
  To evaluate this relationship, the samples will undergo the following analyses: DNA extraction, 16S rRNA amplification, and Illumina MiSeq Sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Cancer Centre; Anna Spreafico, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No